CLINICAL TRIAL: NCT05603130
Title: Diabetes and COVID-19 in Tunisia (CoviDTUN)
Brief Title: Epidemiologic Register on Diabetes and COVID-19 in Tunisia
Status: Completed | Type: Observational
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Other Study IDs: CoviDTUN
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: routinely collected clinical information — medical history, epidemiological characteristics, clinical examination, biological assessment (blood glucose, NFS, CRP, D-dimer,etc...)

SUMMARY:
CoviDTUN is a multicenter observatory set up by a steering committee to determine the presentation and evolution of diabetes in COVID-19 and study its pathogenesis.

The observatory comprises a dataset consisting of routinely collected clinical information anonymously to be entered by the investigator as a participating clinician/researcher.

The study will be an opportunity to understand the relationship between COVID-19 and diabetes, to enrich Tunisian data on diabetic and de novo diabetic patients who have contracted COVID-19 and to evaluate the prognostic severity factors for better management of these patients.

DETAILED DESCRIPTION:
It is a multicentric Tunisian observatory for COVID-19 patients. Confirmed COVID-19 patients, treated on an outpatient basis, in containment centers or hospitalized in COVID-19 units were included retrospectively from March 2020 and had continued prospectively til June 2022. The study had selected eligible patient recorded for inclusion by free practice physicians and hospital physicians. General data, medical history, epidemiological characteristics, clinical examination, biological assessment (blood glucose, NFS, CRP, D-dimer, etc.), clinical course and complications were therefore recorded in a structured and anonymized database. Data collection was carried out by DACIMA Clinical Suite® solution, in accordance with the normative and regulatory provisions in force in the management of health data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 infection confirmed by an evocative clinical picture according to INEAS score or a positive polymerase chain reaction [PCR] test and/or chest CT specific radiological signs and/or a rapid diagnostic antigen test.
* Diabetes known before COVID-19 (known diabetes patient before COVID-19: Diabetic patient before COVID-19: History in medical record and/or presence of antidiabetic therapy and/or HbA1c ≥ 6.5%).

or

- De novo diabetes (the de novo diabetic patient is defined as: Fasting blood glucose ≥ 1.26 g/L (7mmol/L) or postprandial blood glucose ≥ 2g/L (11.1 mmol/L) within 2 weeks of COVID-19 infection, no history of diabetes before the COVID-19 episode)).

Exclusion criteria:

* children
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed COVID-19 patients, treated on an outpatient basis, in containment centers or hospitalized in COVID-19 units.
Sampling Method: Non-Probability Sample
Enrollment: 811 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Effectiveness of patients with COVID-19 who have developed de novo diabetes. | 3 months
  The de novo diabetic patient is defined as follows: Fasting blood glucose ≥ 1.26 g/L (7mmol/L) or postprandial blood glucose ≥ 2g/L (11.1 mmol/L) within 2 weeks of COVID- 19 infection, no history of diabetes before the COVID-19 episode.

SECONDARY OUTCOMES:
Demographic characteristics of diabetic patients | 3 months
  age, weight, gender, BMI, age of diabetes, diabetes treatments, type of diabetes, diabetes complications, comorbidities (hypertension, heart disease, dyslipidemia), vaccination status (number of doses, type of vaccine), associated treatments, hospitalization, evolution (use of respiratory support, cure, death following COVID-19 infection in diabetic and non-diabetic patients).

CONTACTS AND LOCATIONS:
Overall Officials: Faida AJILI, Pr., Principal Investigator — Department of Internal Medicine at the Military Hospital of Tunis
Locations (1):
- Autoimmune diseases research unit UR17DN02, Department of Internal Medicine at the Military Hospital of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No